CLINICAL TRIAL: NCT01998451
Title: The Discovery of the Double Sphincter in Gallbladder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Chengyi Sun, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: GYGDWK-03
Record Dates: First submitted 2013-11-13; First posted 2013-11-28 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Gallstone
Keywords: double sphincter in gallbladder; recurrence rate of gallstones
MeSH Terms: conditions — Gallstones | interventions — ursodoxicoltaurine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double sphincter group (Experimental): patients from double sphincter group all received Tauroursodeoxycholic acid after surgery for 6 months.
  Interventions: Drug: Tauroursodeoxycholic acid
- general gallbladder sphincter group (Other): patients from general gallbladder sphincter group all received Tauroursodeoxycholic acid after surgery for 6 months.
  Interventions: Drug: Tauroursodeoxycholic acid

INTERVENTIONS:
Drug: Tauroursodeoxycholic acid — patients from double sphincter group and general gallbladder sphincter group all received Tauroursodeoxycholic acid after surgery for 6 months.
  Other Names: TUCA

SUMMARY:
We found a new Double sphincter which located in the neck of gallbladder，we supposed it may be related to control pressure of bile duct.Its formation is related to genetic factors.

DETAILED DESCRIPTION:
To contrast the recurrence rate of gallstones between patients with gallbladder double sphincter and patients with general gallbladder sphincter who underwent the treatment of cholecystolithiasis by minimally invasive cholecystolithotomy with gallbladder reservation. Method:Patients with gallbladder double sphincter and patients with general gallbladder sphincter who underwent the treatment of cholecystolithiasis by minimally invasive cholecystolithotomy with gallbladder reservation in The Affiliated Hospital of Guiyang Medical College from May 2012 to December 2015. We collect these patients' bile during surgery.Patients with gallbladder double sphincter as trial group, patients with general gallbladder sphincter as control group.the overall follow-up period is 3 years. Then the investigators statistically analyze improvement of cholecystolithiasis symptoms, thickness of gall bladder wall, the gallbladder function and the rate of the recurrence of cholesterol gallstone in 2 groups.we also analysis of the genetic differences from bile between two groups.

ELIGIBILITY:
Inclusion Criteria:

- people with gallbladder double sphincter

Exclusion Criteria:

- people without gallbladder double sphincter

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The Discovery of The Double Sphincter in Gallbladder | All the patients will be follow-up for an expected average of 3 years.
  The gallbladder of some gallstone patients contain a new Anatomical structure named Double sphincter which located in the middle of gallbladder，we supposed it may be related to the formation of gallstone and pressure of bile duct.Its formation is related to genetic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Chengyi Sun, M.D., Study Chair — The Affiliated Hospital of Guiyang Medial College
Locations (1):
- The Discovery of the Double Sphincter in Gallbladder, Guiyang, Guizhou, China